CLINICAL TRIAL: NCT06194136
Title: Effects of Photobiomodulation on Neuropathic Pain and Sensation Post-mastectomy: a
Brief Title: Photobiomodulation on Neuropathic Pain and Sensation Post-mastectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research team unable to complete study protocol with identified case participant due to participant and research team schedule/factors. Study will not proceed.
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Kim Dao, Assistant Professor, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tufts U
Record Dates: First submitted 2023-10-14; First posted 2024-01-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-04

CONDITIONS: Neuropathic Pain; Sensation Disorders
MeSH Terms: conditions — Neuralgia; Sensation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PBM Intervention (Experimental): Application of commercially-available PBM over the skin of first the right breast and chest tissue and then the left breast and chest tissue, each for 30 seconds in single application. This intervention is to applied once per day, for a total of three times per week, with a minimum of 24 hours between each application.
  Interventions: Device: PBM light therapy

INTERVENTIONS:
Device: PBM light therapy — The PBM machine consists of a dual light emitting diode (LED) cluster array with 105 light diodes within the 660 nanometer (nm) red light wavelength and the 850 nm near-infrared light wavelength. These wavelengths are both within the ranges noted in previous literature for neuropathic pain (1) and are within the World Association for Photobiomodulation (Laser) Therapy (WALT) guidelines for PBM therapy (2). Dosage will be determined according to the following equation: Laser output Power (Watts) x Time (seconds) divided by Beam Area (cm2)= J/cm2 (1). The PBM unit generates energy equal to 115 mW/cm2 with a surface area of 54.6 cm x 17 cm. Thus, for a target power output of 3.45 J, the participant will have a continuous irradiation duration of 30 seconds for each application (1). The participant will be asked to utilize the PBM device on breast tissue post-mastectomy for 30 seconds 3 times per week with at least 24 hours between each session. The duration of treatment will be 6 weeks.

SUMMARY:
The goal of this case study is to examine the effects of Photobiomodulation (PBM) on neuropathic pain and sensation post-mastectomy in one female participant. Neuropathic pain and somatosensation will be primary measures, along with strength, range of motion testing, and measures of quality of life in response to exposure to PBM for 6 weeks.

DETAILED DESCRIPTION:
The goal of this case study is to examine the effects of Photobiomodulation (PBM) on neuropathic pain and sensation post-mastectomy in one female participant.

The main question[s] it aims to answer are:

* Will there be a difference in subjective neuropathic pain reported after application of PBM using red and near-infrared wavelengths?
* If a difference in symptoms is discovered, how many sessions were administered before such difference was noted?
* Will there be an observed difference in sensation assessment after application of PBM using red and near-infrared wavelengths?
* Will there be an observed difference on upper extremity mobility following application of PBM using red and near-infrared wavelengths?
* Will there be a subjective difference in quality-of-life following application of PBM using red and near-infrared wavelengths?

Participants will be asked to participate in:

1. Initial sensation, range of motion, strength, pain, and quality of life assessments.
2. Observation and demonstration of the PBM application with a study investigator present.
3. Application of the PBM device to both sides of the chest over the breast tissue for a total of 30 seconds 3 times a week for 6 weeks in the participant's home environment without a study investigator present.
4. Documentation of pain and skin observation/sensation after each treatment session.
5. Follow-up assessments of sensation, range of motion, strength, pain, and quality of life at the end of week 6 after all PBM treatments have been conducted.
6. Weekly monitoring of pain, and skin observation/sensation during weeks 7-10 in the absence of treatment intervention.
7. Follow-up telephone calls by a study investigator during weeks 7-10.

Researchers will compare pre and post assessment results of sensation, pain, range of motion, strength, and quality of life for any changes as a result of the PBM therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Status-post mastectomy due to clinical diagnosis of breast cancer
* Physician approval for participation in study
* Independent with all mobility
* Independent with cognitive decision-making

Exclusion Criteria:

* Active Malignancy
* Active Infection

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Pain | Up to 10 weeks
  Pain rating on a 0 to 10 scale
Cutaneous Testing using protocol by Cruccu and Truini. (Cruccu G, Truini A. A review of Neuropathic Pain: From Guidelines to Clinical Practice. Pain Ther. 2017;6(Suppl 1):35-42. doi:10.1007/s40122-017-0087-0) | Up to 10 weeks
  Tactile sensation of light touch (Aβ nerve fibers) will be assessed using a cotton ball, pinprick sensation (Aδ nerve fibers) using a wooden cocktail stick, thermal sensation (Aδ and C nerve fibers) using warm and cold objects, and vibration (Aβ nerve fibers) using a tuning fork.
Semmes Weinstein Monofilament Testing | Up to 10 weeks
  Light touch sensation assessment using monofilaments of different diameters

SECONDARY OUTCOMES:
The Quick Dash Outcome Measure | Up to 10 weeks
  Self-rating outcome measure consisting of activity-based and mobility questions using the upper extremity.
Patient-Reported Outcome Measures Information System (PROMIS) 29 + 2 Profile Measure Profile v2.1 | Up to 10 weeks
  Self-rating outcome measure consisting of activity and emotional-based questions pertaining to participation and quality of life in the presence of neuropathic pain.
Range of motion assessment | Up to 10 weeks
  Use of a standard goniometer to measure standard ranges of motion of the upper extremities into shoulder flexion, abduction, internal rotation, and external rotation.
Strength testing (manual muscle testing and dynamometry) | Up to 10 weeks
  Manual muscle testing will consist of manual resistance applied according to a standardized protocol to assess strength of the upper extremities. Dynamometry will be used simultaneously for a numerical/objective representation of strength

CONTACTS AND LOCATIONS:
Overall Officials: Kim D Dao, DPT, Principal Investigator — Tufts University
Locations (1):
- University of St Augustine, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data, including that from subjective and objective assessment measures, will be stored without identifying information, in a shared password-protected drive shared only with the primary and co-investigators as named on this study.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available to the research team up until 6 months after publication.
Access Criteria: Any future studies that wish to mimic the study protocol for research purposes.

REFERENCES:
- [Background] Baron RH, Fey JV, Borgen PI, Stempel MM, Hardick KR, Van Zee KJ. Eighteen sensations after breast cancer surgery: a 5-year comparison of sentinel lymph node biopsy and axillary lymph node dissection. Ann Surg Oncol. 2007 May;14(5):1653-61. doi: 10.1245/s10434-006-9334-z. Epub 2007 Feb 13. PMID 17295084
- [Background] Mustonen L, Vollert J, Rice ASC, Kalso E, Harno H. Sensory profiles in women with neuropathic pain after breast cancer surgery. Breast Cancer Res Treat. 2020 Jul;182(2):305-315. doi: 10.1007/s10549-020-05681-8. Epub 2020 May 27. PMID 32458104
- [Background] Ilhan E, Chee E, Hush J, Moloney N. The prevalence of neuropathic pain is high after treatment for breast cancer: a systematic review. Pain. 2017 Nov;158(11):2082-2091. doi: 10.1097/j.pain.0000000000001004. PMID 28797014
- [Background] Ezzati K, Fekrazad R, Raoufi Z. The Effects of Photobiomodulation Therapy on Post-Surgical Pain. J Lasers Med Sci. 2019 Spring;10(2):79-85. doi: 10.15171/jlms.2019.13. Epub 2019 Feb 25. PMID 31360374
- [Background] Mogahed H, Badawy M, Aziz N. Low-level laser diode on post modified Radical Mastectomy Lymphedema: a randomized controlled trial. J Adv Pharm Res.2020;10(4):105-109.
- [Background] Santiago R, Gomes S, Ozsarfati J, Zitney M. Photobiomodulation for modulation of neuropathic pain and improvement of scar tissue. Scars Burn Heal. 2022 Oct 26;8:20595131221134052. doi: 10.1177/20595131221134052. eCollection 2022 Jan-Dec. PMID 36310679
- [Background] Cialdai F, Landini I, Capaccioli S, Nobili S, Mini E, Lulli M, Monici M. In vitro study on the safety of near infrared laser therapy in its potential application as postmastectomy lymphedema treatment. J Photochem Photobiol B. 2015 Oct;151:285-96. doi: 10.1016/j.jphotobiol.2015.08.003. Epub 2015 Aug 11. PMID 26355716
- [Background] Cruccu G, Truini A. A review of Neuropathic Pain: From Guidelines to Clinical Practice. Pain Ther. 2017 Dec;6(Suppl 1):35-42. doi: 10.1007/s40122-017-0087-0. Epub 2017 Nov 24. PMID 29178033